CLINICAL TRIAL: NCT04122820
Title: Sensitivity of the Search for a Heterophory-Vertical-Labile (HV-Labile) for Ambulatory Screening for Specific Learning Disabilities (SLD) or Developmental Coordination Disorder (DCD).
Brief Title: Ambulatory Screening for Specific Learning Disabilities (SLD) and Developmental Coordination Disorder (DCD).
Acronym: TDys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CNGE IRMG Association (Other)
Collaborators: Scalab CNRS 9193 (Other)
Responsible Party: Principal Investigator, Luc Virlet, Principal Investigator, Scalab CNRS 9193
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CNGEIRMG 0310; 2019-A00416-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-10-05; First posted 2019-10-10 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Specific Developmental Disorders of Speech and Language; Specific Learning Disorder; Dyslexia, Developmental; Developmental Coordination Disorder; Dyspraxia
Keywords: Specific Learning Disorder; Developmental Coordination Disorder; Specific Developmental Disorders of Speech and Language; Dyslexia, Developmental; Dyspraxia
MeSH Terms: conditions — Language; Specific Learning Disorder; Dyslexia; Motor Skills Disorders; Apraxias

STUDY DESIGN:
Intervention Model Description: Comparison of the presence of a specific learning disability, or a Developmental Coordination Disorder, in the case of the presence or absence of referential instability of central origin.
Who Masked: Outcomes Assessor
Masking Description: An adjudication committee to determine the presence or absence of a specific learning disability will be set up, regardless of the presence of a central reference instability.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Presence of HV-Labile (Other): Presence of vertical heterophoria labile with proprioceptive Maddox
  Interventions: Diagnostic Test: Diagnostic of specific learning disabilities or of Developmental Coordination Disorder
- Absence of HV-Labile (Other): Presence of stable vertical heterophoria or stable orthophoria with proprioceptive Maddox
  Interventions: Diagnostic Test: Diagnostic of specific learning disabilities or of Developmental Coordination Disorder

INTERVENTIONS:
Diagnostic Test: Diagnostic of specific learning disabilities or of Developmental Coordination Disorder — Speech therapy assessment, or occupational therapy. In case of pathological disorder, search for a sensory disorder, and therapeutic management. If the pathological disorder persists for more than six months, elimination of a secondary etiology.

SUMMARY:
To evaluate, in primary care, the sensitivity of Heterophory-Vertical-Labile (HV-Labile) in ambulatory screening for Specific Learning Disabilities (SLD) and Developmental Coordination Disorder (DCD). in children aged 8 to 12 years.

DETAILED DESCRIPTION:
General practitioners during a day of professional training on learning disabilities will be trained to perform the proprioceptive Maddox, to search for a HVLabile.

Each trained practitioner will then test at least six children aged 8 to 12 years old in his or her practice, seen at random

250 to 300 physicians will be trained as part of this research

EXPERIMENTAL DESIGN

* Cross-sectional study with prospective recruitment.
* Search for a Vertical Labile Heterophory (HV-Labile).
* Prescription of a standardized speech and language screening assessment for HV-Labile, and in the same number of children without HV-Labile by secondary coupling.
* Delivery of symptomatic questionnaire.
* In case of learning disabilities, the attending physician should look for a possible etiology.
* Adapted speech therapy care for more than six months.
* Speech and language therapy check-up at more than six months.

ELIGIBILITY:
Inclusion Criteria:

The population studied is composed of children:

* from 8 to 12 years old
* seen for any reason for consultation in general practice
* Schooled in an ordinary environment since the Preparatory Course in France
* Francophone parents
* One of whose parents has signed the consent
* Consent of the child
* Social Insured

Exclusion Criteria:

The background and living conditions that may promote secondary learning disabilities, for example:

* Child with a known intellectual disability (Wisc)
* Child in IME (Institut Médico Educatif)
* Child followed in SESSAD (Specialised education service at home)
* Child not knowing how to answer the questions asked
* Child with a known etiology causing learning disabilities (epilepsy, autism spectrum disorder, hearing impairment, visual impairment (deafness, blindness, low vision))
* Child on treatment (antiepileptic, neuroleptic, antidepressant, anxiolytic)
* Child under the care of a psychiatrist,
* Child followed by the CMP (Centre médico-psychologique)
* Child living in an institution,
* Adopted child
* A child whose mother has experienced known depression during the child's early childhood (0-18 months) because it causes attachment disorders, which can impact the child's development, including learning
* Child of a family that has lived through more than two family recompositions
* Child known to be a victim of abuse.
* Out of school child.

To determine the presence of an HV-Labile

* Child with a known visual correction greater than + or- 2 diopters
* Known amblyopic child
* Known strabic child
* Child with no known binocular vision.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the HV-Labile to SLD or DCD | through study completion, an average of 3 year
  Estimated and provided with its 95% confidence interval.

SECONDARY OUTCOMES:
Specificity of the HV-Labile to SLD or DCD | through study completion, an average of 3 year
  Estimated and provided with its 95% confidence interval.
Positive and negative likelihood ratios | through study completion, an average of 3 year
  Estimated and provided with its 95% confidence interval.
Prevalence of children with HV-Labile | through study completion, an average of 3 year
  Estimated and provided with its 95% confidence interval.
Correlation coefficient between the symptomatic proprioceptive questionnaire and the presence of HV-Labile | through study completion, an average of 3 year
  Estimated and provided with its 95% confidence interval.
Positive predictive values | through study completion, an average of 3 year
  Estimated and provided with its 95% confidence interval.
Negative predictive values | through study completion, an average of 3 year
  Estimated and provided with its 95% confidence interval.

OTHER OUTCOMES:
Calculation of results based on a Cut Off at -1.5 standard deviation, or -2 standard deviation, to determine the presence of a SLD or a DCD | through study completion, an average of 3 year
  Estimated and provided with its 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Virlet, Principal Investigator — SCalab CNRS 9193, Lille University
Locations (1):
- Office-based general practioner, Strasbourg, Alsace, France

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Result] Quercia P, Quercia M, Feiss LJ, Allaert F. The distinctive vertical heterophoria of dyslexics. Clin Ophthalmol. 2015 Sep 25;9:1785-97. doi: 10.2147/OPTH.S88497. eCollection 2015. PMID 26445526
- See also: The study undertaken with 100 all-view children shows a strong correlation between the presence of SDP-HV-labile and the presence of specific learning disorders. She encourages us not to neglect the proprioceptive approach in the study of the SLD. — http://www.softal.fr/IMG/pdf/softa-poster-7_avril_14_-virlet-.pdf